CLINICAL TRIAL: NCT02313896
Title: Cirrhosis Readmission Telehealth Project
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor enrollment
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1403013528
Record Dates: First submitted 2014-12-08; First posted 2014-12-10 (Estimated); Last update posted 2016-10-14 (Estimated); Status verified 2016-10

CONDITIONS: Cirrhosis
MeSH Terms: conditions — Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard of Care (No Intervention): Patients recieve standard care. On discharge they receive an information packet about cirrhosis and hepatic encephalopathy. They will continue to follow with their doctor as usual.
- Phone calls (Experimental): On discharge, patients will receive an information package about cirrhosis and hepatic encephalopathy. In addition to regular visits with the doctor, they will receive phone calls from one of our research providers who will be a nurse practitioner, doctor, or physician assistant. In the first 2 weeks after discharge, they will receive phone calls every other day. For the following 10 weeks, they will receive phone calls once a week.
  Interventions: Behavioral: Phone calls

INTERVENTIONS:
Behavioral: Phone calls — Phone calls from medical staff assess confusion of the patient, and recommend immediate changes to dosage of lactulose.
  Arms: Phone calls

SUMMARY:
This is a 2 year research study to study if post discharge phone calls can help lengthen time to hospital readmissions for patients with encephalopathy.

DETAILED DESCRIPTION:
The purpose of this randomized prospective pilot study is to decrease hospital readmissions for patients with hepatic encephalopathy. Patients who were admitted at YNHH with hepatic encephalopathy will be enrolled. Patients will then be randomized to one of two groups upon discharge. The control group will receive usual standard of care for hepatic encephalopathy (encephalopathy education, cirrhosis brochure, stool chart, and routine follow up with their primary care provider and hepatologist). The intervention group will receive usual standard of care as discussed above and phone calls for a 3-month period after their hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* Age of at least 18
* Patients with known cirrhosis
* Current hospitalization for overt hepatic encephalopathy as categorized by West Haven encephalopathy score of 2 or more
* Current hospitalization found no precipitants triggering encephalopathy as determined by the primary team
* Encephalopathy resolved at time of enrollment
* Has a telephone
* Able to obtain medications

Exclusion Criteria:

* Altered mental status unrelated to cirrhosis
* Acute liver failure
* Expectation of liver transplant within 1 month after enrollment
* Chronic kidney disease with Cr > 2 mg/dL
* Respiratory insufficiency:moderate to sever COPD on pulmonary function test
* Electrolyte imbalances not corrected at enrollment
* Sodium less than 125 mmol/L
* Calcium greater than 10mg/dL
* Potassium < 2.5mmol/L
* Unable to give legal consent
* Deafness
* Infection, spontaneous bacterial peritonitis, gastrointestinal bleeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-07; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Hospital Readmission | up to 3 months
  Time to hospital readmission after discharge during the 3 month study period for hepatic encephalopathy

CONTACTS AND LOCATIONS:
Overall Officials: Guadalupe Garcia-Tsao, MD, Principal Investigator — Yale University
Locations (1):
- Yale New Haven Hospital, New Haven, Connecticut, United States